CLINICAL TRIAL: NCT00001884
Title: Specimen Procurement for Individuals With Pulmonary Fibrosis Associated With Rheumatoid Arthritis
Brief Title: Specimen Collection for Individuals With Lung Disease Associated With Rheumatoid Arthritis
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 990068; 99-H-0068
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2007-12-28

CONDITIONS: Pulmonary Fibrosis; Rheumatoid Arthritis
Keywords: Bronchoscopy; Idiopathic Pulmonary Fibrosis; Proteases; Fibroblast Proliferation; Reactive Proteins; Rheumatoid Arthritis; Pulmonary Fibrosis
MeSH Terms: conditions — Pulmonary Fibrosis; Arthritis, Rheumatoid; Idiopathic Pulmonary Fibrosis

SUMMARY:
Pulmonary fibrosis (PF) is a condition in which the lungs of a patient become scarred and fibrous. It has been known to occur in as many as 40% of patients diagnosed with rheumatoid arthritis (RA). The cause of the pulmonary fibrosis in patients with RA is unknown.

Researchers hope to improve their understanding of the disease process involved in PF and RA by analyzing specimens collected by bronchoscopy, lung biopsy, lung transplantation, or autopsy from patients with these conditions.

The purpose of this study is to collect specimens from rheumatoid arthritis patients with and without pulmonary fibrosis as well as patients with pulmonary fibrosis without associated diseases or cause (idiopathic pulmonary fibrosis).

DETAILED DESCRIPTION:
The etiology of pulmonary fibrosis in individuals with rheumatoid arthritis is unknown. Analysis of blood and specimens procured by bronchoscopy, lung biopsy, lung transplantation, or post-mortem examination from patients with this disorder will contribute to our understanding of the pathogenetic mechanisms of pulmonary fibrosis in rheumatoid arthritis. The purpose of this protocol is to obtain blood and specimens by bronchoscopy, lung biopsy, lung transplantation, or post-mortem examination from rheumatoid arthritis patients with and without pulmonary fibrosis, individuals with idiopathic pulmonary fibrosis, and healthy research volunteers.

ELIGIBILITY:
* INCLUSION CRITERIA:

Non-smokers (never smoked or not smoked within the previous 2 years) who are 18 years of age or older with any of the following:

RA with PF (biopsy-proven), or

RA-only, or

Idiopathic PF-only (biopsy-proven), or

Healthy research volunteers by history and indicated tests (individuals without history of chronic cardiopulmonary disorder, collagen vascular disease, or bleeding disorder) matched for age (within 5 years) and gender.

EXCLUSION CRITERIA:

Individuals with any of the following:

Forced expiratory volume in one second (FEV(1)) less than 1L.

Inhalational exposure to fibrogenic fibers or dusts (i.e., asbestos, silica, coal, beryllium).

Chronic cardiopulmonary disorders other than pulmonary fibrosis.

Other collagen vascular disorders (i.e., systemic lupus erythematosus, scleroderma, polymyositis, mixed connective tissue disease).

Non-rheumatoid arthritis.

Viral infections associated with PF (i.e., hepatitis B, hepatitis C, human immunodeficiency virus).

Uncorrectable bleeding diathesis.

Pregnancy or lactation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Start 1999-03-21; Study Completion 2007-12-28

CONTACTS AND LOCATIONS:
Locations (1):
- Boston University, Boston, Massachusetts, United States

REFERENCES:
- [Background] Michalski JP, McCombs CC, Scopelitis E, Biundo JJ Jr, Medsger TA Jr. Alpha 1-antitrypsin phenotypes, including M subtypes, in pulmonary disease associated with rheumatoid arthritis and systemic sclerosis. Arthritis Rheum. 1986 May;29(5):586-91. doi: 10.1002/art.1780290502. PMID 3487321